CLINICAL TRIAL: NCT00117156
Title: A Phase II Study of Fludarabine and Rituximab for the Treatment of Marginal Zone Non-Hodgkin's Lymphoma
Brief Title: Fludarabine and Rituximab for the Treatment of Marginal Zone Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); University of Rochester (Other); Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-294
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma, Non-Hodgkin; MALT Lymphoma
Keywords: Fludarabine; Rituximab; Marginal Zone Lymphoma; MALT lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone | interventions — fludarabine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine and Rituximab (Experimental): Fludarabine:
  25 mg/m2 on days 1-5 of 28 day cycle up to 6 cycles
  Rituximab:
  375 mg/m2 on day 1 of 28 day cycle up to 6 cycles Rituximab dose was split between days 1 and 3 for patients with absolute lymphocyte counts > 10x10^9/L
  Patients received three cycles of therapy followed by re-staging with chest/ abdomen/ pelvic CT scan. Patients with progressive disease discontinued treatment. Patients with stable or responding disease continued therapy for another 3 cycles.
  Interventions: Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine
Drug: Rituximab

SUMMARY:
The purpose of this study is to determine the effectiveness of six cycles of concurrent fludarabine and rituximab in patients with mucosa-associated lymphoid tissue (MALT) lymphoma, marginal zone lymphoma (MZL) or CD5-, CD10-, CD20+ low-grade B cell lymphomas.

DETAILED DESCRIPTION:
Objectives:

Primary

- To estimate the objective response rate.

Secondary

* To assess the safety.
* To describe the progression-free survival at one year.
* To examine the association between clonal cytogenetic abnormalities identified by FISH, and the objective response rate as well as the progression-free survival at one year.

Target enrollment was 30 eligible patients. An 80% objective response rate at 1 month restaging after 6 cycles was considered as evidence of activity in this patient population while 60% was not considered activity. If at least 22 patients achieved objective response the treatment would be considered promising. With 30 eligible patients, the probability of observing this was 0.87 assuming a true rate of 80% and 0.09 assuming a true rate of 60%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed or relapsed MALT, marginal zone lymphoma, or low-grade B cell lymphoproliferative disorder which is CD5-, CD10- and CD20+
* Pathology must be reviewed at Brigham & Women's Hospital, Massachusetts General Hospital, or the University of Rochester James P. Wilmot Cancer Center prior to enrollment
* Documentation of CD20+ status
* Must not be a candidate for local radiotherapy with curative intent
* If gastric MALT, not a candidate for antibiotic therapy with curative intent
* Patients with leukemic phase marginal zone lymphoma are eligible if their absolute lymphocyte count is >10,000 / µl
* Prior treatment with rituximab is permitted, if rituximab induced an objective response which persisted for at least 6 months
* Prior radiotherapy is acceptable
* Measurable disease
* ANC: > 1000/mm3
* Platelets: > 100,000/mm3
* Hemoglobin: > 7 gm/dL
* Adequate renal function as indicated by serum creatinine <= 2 mg/dL.
* Adequate liver function, as indicated by serum total bilirubin <= 2 mg/dL.
* AST or ALT <3x Upper Limit of Normal unless related to primary disease.
* Men and women of reproductive potential must agree to use an acceptable method of birth control during study treatment and for six months after completion of study treatment.
* WHO Performance status </= 2
* Subject has provided written informed consent.

Exclusion Criteria:

* Patients with Waldenstrom's Macroglobulinemia or lymphoplasmacytic lymphoma are excluded
* History of HIV
* Active infection
* Known CNS disease
* Pregnant (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or currently lactating women
* Prior treatment within the last three weeks
* Prior fludarabine
* Positive direct antiglobulin test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-12; Primary Completion 2008-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Rochester Cancer Center, Rochester, New York

REFERENCES:
- [Result] Brown JR, Friedberg JW, Feng Y, Scofield S, Phillips K, Dal Cin P, Joyce R, Takvorian RW, Fisher DC, Fisher RI, Liesveld J, Marquis D, Neuberg D, Freedman AS. A phase 2 study of concurrent fludarabine and rituximab for the treatment of marginal zone lymphomas. Br J Haematol. 2009 Jun;145(6):741-8. doi: 10.1111/j.1365-2141.2009.07677.x. Epub 2009 Mar 30. PMID 19344412

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine and Rituximab: Fludarabine:
  25 mg/m2 on days 1-5 of 28 day cycle up to 6 cycles
  Rituximab:
  375 mg/m2 on day 1 of 28 day cycle up to 6 cycles Rituximab dose was split between days 1 and 3 for patients with absolute lymphocyte counts > 10x10^9/L
  Patients received three cycles of therapy followed by re-staging with chest/ abdomen/ pelvic CT scan. Patients with progressive disease discontinued treatment. Patients with stable or responding disease continued therapy for another 3 cycles.
  Fludarabine
  Rituximab
Period: Overall Study
Arm/Group | Fludarabine and Rituximab
Started | 26
Completed | 15
Not Completed | 11
Not completed — Adverse Event | 9
Not completed — Physician Decision | 1
Not completed — Trt for Pre-Exist Second Primary | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine and Rituximab
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 63.7 [31.4 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 26
Histology [Number; unit: participants]
  Nodal MZL | 14
  MALT | 8
  Splenic MZL | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is defined as the proportion of patients who achieve complete remission (CR), complete remission/unconfirmed (CRu) or partial remission (PR) based on Cheson criteria (1999).
Time Frame: Assessed after three- and six-cycles of therapy.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Fludarabine and Rituximab
Number analyzed (Participants) | 26
proportion of patients | .85 [.65 to .96]

2. Secondary Outcome: 3.1-Year Progression-Free Survival
Description: 3.1-year progression-free survival is the probability of patients remaining alive and progression-free at 3.1 years from study entry estimated using Kaplan-Meier methods. Disease progression was assessed per Cheson criteria (1999).
Time Frame: Assessed after 3- and 6-cycles of therapy, every 6 months for 2 years and then annually up to 4 years
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Fludarabine and Rituximab
Number analyzed (Participants) | 26
probability | 0.795 [0.634 to 0.956]

3. Secondary Outcome: 3.1-Year Overall Survival
Description: 3.1-year overall survival is the probability of patients remaining alive 3.1 years from study entry.
Time Frame: Assessed after 3- and 6-cycles of therapy, every 6 months for 2 years and then annually up to 4 years
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Fludarabine and Rituximab
Number analyzed (Participants) | 26
probability | 0.874 [0.74 to .99]

4. Post Hoc Outcome: Delayed Bone Marrow Toxicity Rate
Description: Delayed bone marrow toxicity rate is the proportion of patients who experienced significant bone marrow toxicity defined as aplastic anemia or myelodysplastic syndromes (MDS) after completing therapy.
Time Frame: Assessed after therapy completion incidentally or at a minimum every 6 months for 2 years and then annually up to 4 years.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Fludarabine and Rituximab
Number analyzed (Participants) | 26
proportion of patients | 0.154 [0.043 to 0.349]

5. Post Hoc Outcome: Delayed Pneumonia Toxicity Rate
Description: Delayed pneumonia toxicity rate is the proportion of patients who experienced significant pneumonia toxicity defined as nocardia or pneumocystis jiroveci after completing therapy.
Time Frame: as for outcome 4
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Fludarabine and Rituximab
Number analyzed (Participants) | 26
proportion of patients | 0.115 [0.024 to 0.301]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment.
Description: Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3.
  Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Fludarabine and Rituximab
Serious Adverse Events (participants affected / at risk) | 20/26
Other Adverse Events (participants affected / at risk) | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine and Rituximab (N=26)
Hemoglobin (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever w/o neutropenia (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Leukocytes (Investigations) | 11
Neutrophils (Investigations) | 15
Platelets (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine and Rituximab (N=26)
Hemoglobin (Blood and lymphatic system disorders) | 15
Sinus tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 16
Fever w/o neutropenia (General disorders) | 5
Rigors/chills (General disorders) | 3
Constitutional, other (General disorders) | 1
Edema limb (General disorders) | 1
Allergic reaction (Immune system disorders) | 5
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Leukocytes (Investigations) | 9
Neutrophils (Investigations) | 4
Platelets (Investigations) | 6
Alkaline phosphatase (Investigations) | 1
ALT, SGPT (Investigations) | 2
AST, SGOT (Investigations) | 2
Bilirubin (Investigations) | 2
Creatinine (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 1
Neurologic-other (Nervous system disorders) | 2
Head/headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No